CLINICAL TRIAL: NCT01618929
Title: Phase 4 Study of Effects of Montelukast Treatment on Allergic Inflammation in Children With and Without Food Allergy, Single Centered, Randomised, Double Blind, Placebo Controlled Parallel Group Cross-over Study
Brief Title: Effects of Montelukast in Asthmatic Children With and Without Food Allergy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hacettepe University (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Cansin Sackesen, Associate Professor, Hacettepe University
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MISP Protocol 1.0
Record Dates: First submitted 2012-06-12; First posted 2012-06-13 (Estimated); Last update posted 2017-08-14 (Actual); Status verified 2017-08

CONDITIONS: Bronchial Asthma; Food Allergy; Children
Keywords: Food allergy; Asthma; Children; Montelukast; Inflammation
MeSH Terms: conditions — Asthma; Food Hypersensitivity; Inflammation | interventions — montelukast

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- asthma with food allergy (Active Comparator): The study will be performed in 2 groups of patients (Patients with and without food allergy) parallel to each other at the same time and within each group the patients will take montelukast and placebo (one after another in a double-blind design).
  Interventions: Drug: Montelukast
- asthma without food allergy (Active Comparator): The study will be performed in 2 groups of patients (Patients with and without food allergy) parallel to each other at the same time and within each group the patients will take montelukast and placebo (one after another in a double-blind design)
  Interventions: Drug: Montelukast

INTERVENTIONS:
Drug: Montelukast — Placebo and montelukast (5 mg for 6-14 years of age and 10 mg for 14-18 years of age once a day) will be given following one another in 4 weeks periods including a 2 weeks wash-out period in between in a cross over design.
  Other Names: Singulair 5 mg tablets; Singulair 10 mg tablets; Placebo 5 mg tablets; Placebo 10 mg tablets

SUMMARY:
* To search the effects of montelukast on the airway inflammation including FEV1%, FEV1%/FVC, the provocholine® (methacoline chloride powder for inhalation) challenge tests, the leukotriene levels in the exhaled breath condensate in asthmatic children with and without food allergy aged 6-18 years old.
* To define the patient groups with good response to montelukast and to define the parameters which predict the good response.

DETAILED DESCRIPTION:
The aim of this analysis is to determine whether the children with food allergy may have more eosinophilic inflammation in the airways (as measured by FENO) or they may have Cysteinyl leukotrienes based inflammation in the airways that will be shown by high levels of Cys LT and low levels of lipoxin in the exhaled breath condensate. Our suggestion is that a special pattern of inflammation may be seen in asthmatics with food allergy because of their strong atopic march history and then we aimed to test if montelukast is more effective in children when the ratio of Cysteinyl LT inflammation is high relative to FENO (eosinophilic inflammation). This study will be the first to evaluate the effect of montelukast regarding the synthesis of Cys leukotrienes, lipoxin and FENO that will be measured from exhaled breath condensate, which is the mirror of the local inflammation in the airways in asthmatic children with atopy (food allergy). As we mentioned above another factor that we are planning to analyze is the ratio of Cys leukotriene to lipoxin, which is the natural antagonist of LT. This study will determine the ratio of Cyst LT to lipoxin and Cyst LT to FENO in the exhaled breath condensate and then there will be an analysis to see the correlation of these inflammatory markers with montelukast related changes on FEV1%, FEV1%/FVC.

ELIGIBILITY:
Inclusion Criteria:

* Physician diagnosed asthma (12% reversibility on spirometry test or positive response to provocholine® provocation test).
* Mild to moderate asthmatic children. Asthmatic children with pre-budesonide FEV1/FVC ≥ 80% will be included.
* At least one food allergy confirmed by specific IgE level or skin prick test positivity and a relevant clinical history or open challenge test with food.
* Aged between 6-18 years old.
* Acceptance of involvement in the study and signed informed consent (Both patients and one of the parents)

Exclusion Criteria:

* Who does not sign the informed consent.
* Severe asthmatic children
* Any lung disease except asthma (i.e. cystic fibrosis, bronchiectasia, primary ciliary dyskinesia).
* Any systemic disease except allergic rhinitis and atopic dermatitis
* Follow-up in intensive care unit or intubation for asthma exacerbation within one year.
* Attendance to emergency room or hospital admission within 3 months for asthma exacerbation
* Systemic steroid usage within 3 months
* Upper airway infection within one month.
* Psychiatric or psychosocial problems
* Poor compliance to asthma treatment protocol
* Any condition contra-indicated for montelukast usage
* To be aware of the name of the drug either patient or study staff during the study period.
* Worsening of the clinical condition during run-in period.
* Pregnancy or breast feeding

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 113 (Actual)
Dates: Start 2013-03; Primary Completion 2015-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
the difference in FEV1% between two arms. | 10 weeks
  The asthmatic children with and without food allergy will be given placebo and montelukast following one another in a cross over design. The study will be performed in 2 groups of patients (Patients with and without food allergy) parallel to each other at the same time and within each group the patients will take montelukast and placebo. A total of 5 spirometry tests (At the beginning and end of run-in periods, at the beginning of cross-over period, at the end of wash-out period and at the end of the study) will be done and forced expiratory volume in one second (FEV1) will be evaluated.

SECONDARY OUTCOMES:
Exhaled breath condensate | 14 weeks
  It will be collected 4 times during the study period (At the beginning and at the end of drug and placebo usage periods.)Cysteinyl leukotrienes, Prostaglandin D2, lipoxin levels will be measured in the exhaled breathe condensate
Fractional exhaled Nitric Oxide | 14 weeks
  It's measurement will be done 4 times during the study period (At the beginning and at the end of drug and placebo usage periods.) (See flow chart).
asthma control test | 14 weeks
bronchial hyperreactivity | 14 weeks
  In order to document the level of bronchial hyperreactivity of the patients, the provocholine (methacholine chloride powder for inhalation) provocation tests will be performed 4 times (At the beginning and at the end of drug and placebo usage periods)

CONTACTS AND LOCATIONS:
Overall Officials: Cansin Sackesen, Assoc Prof, Study Chair — Hacettepe University; Umit M Sahiner, MD, Principal Investigator — Hacettepe University; Betul Buyuktiryaki, MD, fellow, Principal Investigator — Hacettepe University; Ozlem Cavkaytar, MD, fellow, Principal Investigator — Hacettepe University; Ebru Arikyılmaz, MD, fellow, Principal Investigator — Hacettepe University; Ayfer Tuncer, Professor, Principal Investigator — Hacettepe University; Ozge U Soyer, Assist Prof, Principal Investigator — Hacettepe University
Locations (1):
- Cansin Sackesen, Ankara, Turkey (Türkiye)

REFERENCES:
- [Background] Szefler SJ, Phillips BR, Martinez FD, Chinchilli VM, Lemanske RF, Strunk RC, Zeiger RS, Larsen G, Spahn JD, Bacharier LB, Bloomberg GR, Guilbert TW, Heldt G, Morgan WJ, Moss MH, Sorkness CA, Taussig LM. Characterization of within-subject responses to fluticasone and montelukast in childhood asthma. J Allergy Clin Immunol. 2005 Feb;115(2):233-42. doi: 10.1016/j.jaci.2004.11.014. PMID 15696076
- [Background] Rabinovitch N, Graber NJ, Chinchilli VM, Sorkness CA, Zeiger RS, Strunk RC, Bacharier LB, Martinez FD, Szefler SJ; Childhood Asthma Research and Education Network of the National Heart, Lung, and Blood Institute. Urinary leukotriene E4/exhaled nitric oxide ratio and montelukast response in childhood asthma. J Allergy Clin Immunol. 2010 Sep;126(3):545-51.e1-4. doi: 10.1016/j.jaci.2010.07.008. PMID 20816189